CLINICAL TRIAL: NCT02577198
Title: Implementing an Evidence-based Computerized Decision Support System Linked to Electronic Health Records to Improve Patient Care in a General Hospital
Brief Title: Computerized Decision Support System Linked to Electronic Health Records to Improve Patient Care in a General Hospital
Acronym: CODES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Collaborators: University of Milan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: C41J11000110008
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-10

CONDITIONS: Physician's Role

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Electronic Health Records with computerised decision support system activated Medilogy Decision Support System (MediDSS)
  Interventions: Other: Medilogy Decision Support System (MediDSS)
- Control (Other): Electronic Health Records with computerised decision support system silenced Medilogy Decision Support System (MediDSS) silenced
  Interventions: Other: Medilogy Decision Support System (MediDSS)

INTERVENTIONS:
Other: Medilogy Decision Support System (MediDSS) — Italian translation of Evidence-Based Medicine electronic Decision Support (EBMeDS), a set of rules (scripts) based on Evidence Based Medicine guidelines and applied to structured health data. MediDSS further includes knowledge from Swedish, Finnish, INteraction X-referencing (SFINX), a drug-drug interaction database containing concise evidence-based information of about 18,000 drug interactions and adverse events. MediDSS is integrated with local reminders.

SUMMARY:
Computerized decision support systems (CDSSs) are information technology-based software that provide health professionals with actionable, patient-specific recommendations or guidelines for disease diagnosis, treatment, and management at the point-of-care. CDSSs may be integrated with patient electronic health records (EHRs) and evidence-based knowledge.

DETAILED DESCRIPTION:
The investigators designed a pragmatic randomized controlled trial to evaluate the effectiveness of patient-specific, point-of-care reminders on clinical practice and the quality of care. The investigators hypothesize that these reminders can increase clinician adherence to guidelines and, eventually, improve the quality of care offered to hospitalized patients. The results of the investigators study will contribute to the current understanding of the effectiveness of CDSSs in primary care and hospital settings.

ELIGIBILITY:
Inclusion Criteria:

All of the patients admitted into the internal medicine departments of the Azienda Ospedaliera di Desio e Vimercate during the study period.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6479 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Resolution rates | 12 months
  Rate at which the medical problems, which are detected by the MediDSS software and reported through the reminders, are resolved (resolution rates).

SECONDARY OUTCOMES:
in-hospital mortality | 12 months
length of hospital stay | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Lorenzo Moja, MD, PhD, Principal Investigator — Unità di Epidemiologia Clinica, IRCCS Istituto Ortopedico Galeazzi, Milano
Locations (1):
- Ospedale di Vimercate, Vimercate, Lombardy, Italy

REFERENCES:
- [Background] Moja L, Kwag KH, Lytras T, Bertizzolo L, Brandt L, Pecoraro V, Rigon G, Vaona A, Ruggiero F, Mangia M, Iorio A, Kunnamo I, Bonovas S. Effectiveness of computerized decision support systems linked to electronic health records: a systematic review and meta-analysis. Am J Public Health. 2014 Dec;104(12):e12-22. doi: 10.2105/AJPH.2014.302164. Epub 2014 Oct 16. PMID 25322302
- [Background] Moja L, Liberati EG, Galuppo L, Gorli M, Maraldi M, Nanni O, Rigon G, Ruggieri P, Ruggiero F, Scaratti G, Vaona A, Kwag KH. Barriers and facilitators to the uptake of computerized clinical decision support systems in specialty hospitals: protocol for a qualitative cross-sectional study. Implement Sci. 2014 Aug 28;9:105. doi: 10.1186/s13012-014-0105-0. PMID 25163794
- [Background] Liberati EG, Galuppo L, Gorli M, Maraldi M, Ruggiero F, Capobussi M, Banzi R, Kwag K, Scaratti G, Nanni O, Ruggieri P, Polo Friz H, Cimminiello C, Bosio M, Mangia M, Moja L. [Barriers and facilitators to the implementation of computerized decision support systems in Italian hospitals: a grounded theory study]. Recenti Prog Med. 2015 Apr;106(4):180-91. doi: 10.1701/1830.20032. Italian. PMID 25959891
- [Background] Moja L, Polo Friz H, Capobussi M, Kwag K, Banzi R, Ruggiero F, Gonzalez-Lorenzo M, Liberati EG, Mangia M, Nyberg P, Kunnamo I, Cimminiello C, Vighi G, Grimshaw J, Bonovas S. Implementing an evidence-based computerized decision support system to improve patient care in a general hospital: the CODES study protocol for a randomized controlled trial. Implement Sci. 2016 Jul 7;11(1):89. doi: 10.1186/s13012-016-0455-x. PMID 27389248
- [Derived] Moja L, Polo Friz H, Capobussi M, Kwag K, Banzi R, Ruggiero F, Gonzalez-Lorenzo M, Liberati EG, Mangia M, Nyberg P, Kunnamo I, Cimminiello C, Vighi G, Grimshaw JM, Delgrossi G, Bonovas S. Effectiveness of a Hospital-Based Computerized Decision Support System on Clinician Recommendations and Patient Outcomes: A Randomized Clinical Trial. JAMA Netw Open. 2019 Dec 2;2(12):e1917094. doi: 10.1001/jamanetworkopen.2019.17094. PMID 31825499